CLINICAL TRIAL: NCT01820169
Title: Study on Improvement of Blood Glucose Control in Patients With Diabetes Type 2 Using SMBG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 2 patients screened but none of them were enrolled.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001551
Record Dates: First submitted 2013-03-11; First posted 2013-03-28 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

ARMS (1):
- Single arm (Experimental)
  Interventions: Device: ;Accu-Chek Compact Plus LCM bulk Japan

INTERVENTIONS:
Device: ;Accu-Chek Compact Plus LCM bulk Japan — HbA1c would be changed by more careful control in blood glucose with SMBG.

SUMMARY:
This clinical study is to determine if the use of structured testing, which is a blood glucose monitoring, via the Accu-Chek 360° View blood glucose analysis tool has a positive effect on the subjects overall glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Age:= and >20 years. 2. Intend to paticipate in this study after education of structured testing. 3.HbA1c:= and >7.5% in the recect 2 months.

Exclusion Criteria:

1.Pregancy. 2. Heavy complication 3. judged unsuitable by doctor

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improvement in HbA1c in 6 months | 6 months

SECONDARY OUTCOMES:
1. Comparison with historical control in HbA1c change. | Baseline to 6 months
2. Change in blood gulucose. | Baseline to 6 months
3. Change in BMI. | Baseline to 6 months
4. Occurance of sever hypoglycemia. | Baseline to 6 months
5. Doctor's opinion for Accu-Chek 360° View. | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Sakane, Principal Investigator — National organization Hospital Kyoto Medical Center
Locations (1):
- Kyoto, Japan